CLINICAL TRIAL: NCT03227991
Title: Safety Planning Intervention to Reduce Short Term Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: University of Pennsylvania (Other); University of Massachusetts, Worcester (Other); Columbia University (Other); American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Beth Brodsky, Associate Director, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7383
Record Dates: First submitted 2016-12-15; First posted 2017-07-24 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Suicide, Attempted
Keywords: Suicide
MeSH Terms: conditions — Suicide, Attempted; Suicide | interventions — Risk Factors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Planning Intervention (Active Comparator): SPI is a personalized approach that focuses on early identification of warning signs and execution of systematic steps to manage suicidal thoughts, created collaboratively by the patient and clinician.
  Interventions: Behavioral: Safety Planning Intervention
- Risk factors and Warning signs (Active Comparator): Patients will receive a generic suicide risk factors and warning signs information handout.
  Interventions: Behavioral: Risk factors and Warning signs

INTERVENTIONS:
Behavioral: Safety Planning Intervention — The Safety Planning Intervention is a protocol driven, brief suicide prevention strategy that is a good fit for acute care settings. It involves a clinician working collaboratively with the patient to build a personalized safety plan that is documented using a templated paper form and includes warning sign identification, means restriction and personalized strategies to deescalate a suicide crisis.
  Other Names: SPI
  Arms: Safety Planning Intervention
Behavioral: Risk factors and Warning signs — Printed information sheet listing suicide risk factors and crisis hotlines
  Other Names: RWI
  Arms: Risk factors and Warning signs

SUMMARY:
This study will determine the efficacy of Safety Planning Intervention (SPI) compared to receiving risk factors and warning sign information (RWI) in recent suicide attempters during the 6 months following an acute care visit on: (1) suicidal behaviors; (2) mental health/substance use treatment engagement; (3) suicide-related coping strategies; (4) suicidal ideation; and (5) use of means restriction.

DETAILED DESCRIPTION:
There is a pressing need for improved acute care setting suicide prevention interventions. The Safety Planning Intervention (SPI) is a protocol driven, brief suicide prevention strategy that is a good fit for acute care settings (i.e., emergency departments (ED) and inpatient units). The SPI involves a clinician working collaboratively with the patient to build a personalized safety plan that is documented using a templated paper form and includes warning sign identification, means restriction and personalized strategies to deescalate a suicide crisis. It is easy to learn and administer, acceptable to patients, brief, firmly rooted in an empirical base and has preliminary studies supporting its feasibility and potential to impact patient outcomes, including suicidal behavior and treatment engagement. However, while it is being adopted widely, it lacks a randomized controlled trial (RCT) to definitively determine its efficacy. The purpose of this study to conduct a randomized control trial of the Safety Planning Intervention (SPI) compared with receiving risk factors and warning sign information (RWI) in acute care settings.

All participants in this study will complete some baseline assessments, following which they will be randomly assigned to one of two study conditions: Safety Plan Intervention (SPI) or receiving risk factors and warning sign information (RWI). If assigned to SPI, participants will receive the assigned intervention by the research clinician. They will receive a paper copy of their safety plan while in the ED or on the inpatient unit and a back-up copy will be sent approximately 1 week after discharge to participants. For RWI participants, ED and inpatient unit care will be delivered as usual, with the addition of a printed information sheet listing suicide risk factors and crisis hotlines. In addition to the baseline assessment, multi-method outcome assessment will be conducted at 1, 3, and 6 months. This will include telephone evaluations by a blinded assessor (not the research clinician), medical record review, and vital statistics registry review.

ELIGIBILITY:
Inclusion Criteria:

1. Presented for an acute care visit within 8 weeks of a suicide attempt, interrupted or aborted attempt, or suicidal ideation with intent and plan within 4 weeks.
2. Are 18 years of age or older
3. Able to speak and read English
4. Able to understand the nature of the study, provide written informed consent, and complete study procedures
5. Have been evaluated by a health care professional who provides permission for research staff to approach the patient.

Exclusion Criteria:

1. Under 18 years of age
2. Cannot speak or read English
3. Unable to understand the nature of the study, provide written informed consent, or complete study procedures
4. Unable or unwilling to provide a personal phone number for follow up purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Suicide, attempted and suicide | 1 month
  As measured by the Columbia Suicide Severity Rating Scale (C-SSRS); responses are yes-no with yes more severe
Suicide, attempted and suicide | 3 months
  As measured by the Columbia Suicide Severity Rating Scale (C-SSRS); responses are yes-no with yes more severe
Suicide, attempted and suicide | 6 months
  As measured by the Columbia Suicide Severity Rating Scale (C-SSRS); responses are yes-no with yes more severe

SECONDARY OUTCOMES:
Suicide, attempted, aborted, interrupted attempt or preparatory suicidal behavior | 1 month
  As measured by the Columbia Suicide Severity Rating Scale (C-SSRS); responses are yes-no with yes more severe
Suicide, attempted, aborted, interrupted attempt or preparatory suicidal behavior | 3 months
  As measured by the Columbia Suicide Severity Rating Scale (C-SSRS); responses are yes-no with yes more severe
Suicide, attempted, aborted, interrupted attempt or preparatory suicidal behavior | 6 months
  As measured by the Columbia Suicide Severity Rating Scale (C-SSRS); responses are yes-no with yes more severe
Means restriction | 1 month
  As measured by patient report about reducing access to lethal means
Means restriction | 3 months
  As measured by patient report about reducing access to lethal means
Means restriction | 6 months
  As measured by patient report about reducing access to lethal means
Suicide related coping | 1 month
  As measured by the total score on the Suicide-Related Coping Measure, a scale developed by Stanley, Brown and Holloway (2010). The scale is a 21 item self-report measure using a Likert scale. Examples of items are: "I am at the mercy of my suicidal thoughts." and "I have several things I can do to get through a suicidal crisis." The scale has high in internal reliability (Cronbach's alpha = .88), and, as predicted, moderate convergent validity with help-seeking attitudes (r = .47) and divergent validity with a pain measure (r= -.31). It is also sensitive to change (t(65) = 6.8, p < .001).
Suicide related coping | 3 months
  As measured by the total score on the Suicide-Related Coping Measure, a scale developed by Stanley, Brown and Holloway (2010). The scale is a 21 item self-report measure using a Likert scale. Examples of items are: "I am at the mercy of my suicidal thoughts." and "I have several things I can do to get through a suicidal crisis." The scale has high in internal reliability (Cronbach's alpha = .88), and, as predicted, moderate convergent validity with help-seeking attitudes (r = .47) and divergent validity with a pain measure (r= -.31). It is also sensitive to change (t(65) = 6.8, p < .001).
Suicide related coping | 6 months
  As measured by the total score on the Suicide-Related Coping Measure, a scale developed by Stanley, Brown and Holloway (2010). The scale is a 21 item self-report measure using a Likert scale. Examples of items are: "I am at the mercy of my suicidal thoughts." and "I have several things I can do to get through a suicidal crisis." The scale has high in internal reliability (Cronbach's alpha = .88), and, as predicted, moderate convergent validity with help-seeking attitudes (r = .47) and divergent validity with a pain measure (r= -.31). It is also sensitive to change (t(65) = 6.8, p < .001).
Treatment engagement | 1 month
  As measured by attending one of more mental health/substance abuse treatment appointments
Treatment engagement | 3 months
  As measured by attending one of more mental health/substance abuse treatment appointments
Treatment engagement | 6 months
  As measured by attending one of more mental health/substance abuse treatment appointments
Suicidal ideation intensity | 1 month
  As measured by the Columbia Suicide Severity Rating Scale (CSSRS) on a scale from 1-5
Suicidal ideation intensity | 3 months
  As measured by the Columbia Suicide Severity Rating Scale (CSSRS) on a scale from 1-5
Suicidal ideation intensity | 6 months
  As measured by the Columbia Suicide Severity Rating Scale (CSSRS) on a scale from 1-5
Suicidal ideation severity | 1 month
  As measured by the Columbia Suicide Severity Rating Scale (CSSRS) on a scale from 2-25 with higher scores more severe
Suicidal ideation severity | 3 months
  As measured by the Columbia Suicide Severity Rating Scale (CSSRS) on a scale from 2-25 with higher scores more severe
Suicidal ideation severity | 6 months
  As measured by the Columbia Suicide Severity Rating Scale (CSSRS) on a scale from 2-25 with higher scores more severe

CONTACTS AND LOCATIONS:
Overall Officials: Barbara H Stanley, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (3):
- United States (3):
  - University of Massachusetts, Worcester, Massachusetts
  - New York State Psychiatric Institute, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boudreaux ED, Stanley B, Green KL, Galfalvy H, Brown GK. A randomized, controlled trial of the safety planning intervention: Research design and methods. Contemp Clin Trials. 2021 Apr;103:106291. doi: 10.1016/j.cct.2021.106291. Epub 2021 Jan 27. PMID 33515785